CLINICAL TRIAL: NCT05250622
Title: OrthoEvidence Trial Assessing Japanese Knowledge Updates : Trial of Knowledge Translation Among Japanese Surgeons
Brief Title: OrthoEvidence Trial Assessing Japanese Knowledge Updates
Acronym: OTAKU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Japanese Society for Fracture Repair (Unknown); OrthoEvidence (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 13493
Record Dates: First submitted 2022-01-31; First posted 2022-02-22 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Healthy Volunteer
Keywords: Surveys and Questionnaires; Clinical Competence; Orthopedics; Attitude of Health Personnel; Evidence-based medicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Japanese group (Experimental): Participants who will receive Japanese-translated version of evidence summaries
  Interventions: Other: Japanese-translated evidence summaries (Advanced Clinical Evidence report from OrthoEvidence)
- English group (Active Comparator): Participants who will receive English version of evidence summaries
  Interventions: Other: English evidence summaries (Advanced Clinical Evidence report from OrthoEvidence)

INTERVENTIONS:
Other: Japanese-translated evidence summaries (Advanced Clinical Evidence report from OrthoEvidence) — Participants will receive emails with the link to Japanese-translated version of evidence summaries.
  Arms: Japanese group
Other: English evidence summaries (Advanced Clinical Evidence report from OrthoEvidence) — Participants will receive emails with the link to English version of evidence summaries.
  Arms: English group

SUMMARY:
The purpose of this randomized controlled trial is to clarify whether providing translated evidence summary (Advanced Clinical Evidence (ACE) reports from OrthoEvidence) will increase the access to the summary compared to providing the original version of evidence summary among Japanese orthopaedic surgeons

DETAILED DESCRIPTION:
The investigators will conduct the survey regarding baseline characteristics, barriers and familiality to evidence-based medicine by online. After the survey, the participants will be randomly assigned to receive either the original version of ACE reports or Japanese version of ACE reports. The pdf of each ACE report will be provided to the participants through an email link. Twenty reports will be sent over 4 weeks period. After that, the investigators will conduct another survey regarding the reports.

ELIGIBILITY:
Inclusion Criteria:

1. Member of Japanese Society for Fracture Repair (JSFR)
2. Spend at least 20% of their time in clinical practice
3. Non-native speaker of English
4. Has regular access to internet
5. Prefer to read Japanese-translated material, if there are both translated and English version of the same material.

Exclusion Criteria:

We will exclude surgeons who cannot provide informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Number of access to evidence summaries | Four weeks (28 days) after the commencement of the trial
  Total number of access to evidence summaries

SECONDARY OUTCOMES:
Self-rated score of understanding the contents of the provided materials | Within four weeks after the end of intervention
  Five-point Likert scale in understanding the contents of provided materials, evaluated by the participants (higher scores means better outcome)
Self-rated score in changing their practice based on the contents of the materials | Within four weeks after the end of intervention
  Five-point Likert scale in changing their practice based on the contents of the materials evaluated by the participants (higher scores means better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Madden, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sprague S, Smith C, Bhandari M. OrthoEvidence: A Clinical Resource for Evidence-Based Orthopedics. Orthop Rev (Pavia). 2015 Jun 3;7(2):5762. doi: 10.4081/or.2015.5762. eCollection 2015 Jun 3. PMID 26330990
- [Background] Poolman RW, Sierevelt IN, Farrokhyar F, Mazel JA, Blankevoort L, Bhandari M. Perceptions and competence in evidence-based medicine: Are surgeons getting better? A questionnaire survey of members of the Dutch Orthopaedic Association. J Bone Joint Surg Am. 2007 Jan;89(1):206-15. doi: 10.2106/JBJS.F.00633. PMID 17200328
- [Background] Dahm P, Poolman RW, Bhandari M, Fesperman SF, Baum J, Kosiak B, Carrick T, Preminger GM; American Urological Association Membership. Perceptions and competence in evidence-based medicine: a survey of the American Urological Association Membership. J Urol. 2009 Feb;181(2):767-77. doi: 10.1016/j.juro.2008.10.031. Epub 2008 Dec 16. PMID 19091333